CLINICAL TRIAL: NCT05158153
Title: Outpatient Recovery From Acute Kidney Injury Requiring Dialysis
Acronym: ORKID
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inadequate recruitment
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-33602
Record Dates: First submitted 2021-11-19; First posted 2021-12-15 (Actual); Results first posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-04

CONDITIONS: Acute Kidney Injury; Dialysis Hypotension
Keywords: Dialysis-requiring Acute Kidney Injury; Renal Recovery
MeSH Terms: conditions — Acute Kidney Injury | interventions — Furosemide

STUDY DESIGN:
Intervention Model Description: This is a single-center (multi-clinic), non-randomized pilot study to investigate the feasibility, tolerability, and safety of a bundled intervention (cooled dialysate, high sodium dialysate, high dose diuretics, high ultrafiltration hold threshold, active dialysis weaning) designed to foster recovery from acute kidney injury requiring dialysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ORKID Bundled Intervention (Experimental)
  Interventions: Other: ORKID Bundled Intervention; Drug: Furosemide

INTERVENTIONS:
Other: ORKID Bundled Intervention — During the 90-day study period, participants will be prescribed outpatient hemodialysis with cooled dialysate (35-36°C), high sodium dialysate (145 mmol/L), a high ultrafiltration hold threshold (systolic blood pressure > 110 mmHg; ultrafiltration hold threshold will not be applied in participants with baseline systolic blood pressure < 120 mmHg), and high dose diuretics (160 mg oral furosemide twice daily) to be taken every day at home will also be prescribed. Dialysis will be weaned according to an active weaning protocol.
Drug: Furosemide — 160 mg oral furosemide twice daily to be taken every day at home

SUMMARY:
There are currently no therapies to improve the chances of recovering enough kidney function to come off of dialysis after severe acute kidney injury. It is not known if current routine outpatient dialysis treatments are optimized to maximize the chances of recovery. The purpose of this pilot study is to see if we can feasibly and safely provide several changes to the way that dialysis is provided in outpatient dialysis centers which may improve the chances of recovery.

ELIGIBILITY:
Inclusion Criteria:

* AKI-D (acute kidney injury requiring dialysis), attributed at least in part to acute tubular necrosis by clinical nephrology team
* Age ≥ 18 years
* Pre-hospitalization eGFR ≥ 15 mL/min/1.73m2
* Being discharged to a participating outpatient dialysis unit (within 30 miles of UCSF)

Exclusion Criteria:

* Known loop diuretic allergy/intolerance
* Dialysis duration > 3 months
* Pregnant
* Prisoner
* Unable to consent
* Clinical team declines to allow approach for study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian McCoy, MD, MS, Principal Investigator — University of California, San Franisco; Chi-yuan Hsu, MD, MSc, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ORKID Bundled Intervention
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ORKID Bundled Intervention
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Race/Ethnicity | NA — Only 1 participant was enrolled in this study, due to the possibility of identification, data will not be presented.

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Who Received the Dialysate Temperature, Dialysate Sodium Concentration, Diuretic Dose, and Ultrafiltration Hold Threshold That Was Ordered at Least Once in the First Two Weeks of Treatment.
Description: Feasibility
Time Frame: First two weeks of study intervention
Population: Only 1 participant was enrolled in this study, due to the possibility of identification, data will not be presented.
Arm/Group | ORKID Bundled Intervention
Number analyzed (Participants) | 0

2. Secondary Outcome: The Proportion of Enrolled Patients Completing the 90-day Study Still Continuing Each Intervention.
Description: Tolerability
Time Frame: Study day 90
Population: Only 1 participant was enrolled in this study, due to the possibility of identification, data will not be presented.
Arm/Group | ORKID Bundled Intervention
Number analyzed (Participants) | 0

3. Secondary Outcome: Incidence of Adverse Events; Both Serious and Non-serious Adverse Events Will be Monitored Including Electrolyte Abnormalities, Emergent Dialysis Treatments, and Hospitalizations.
Description: Safety
Time Frame: Study day 90
Population: Only 1 participant was enrolled in this study, due to the possibility of identification, data will not be presented.
Arm/Group | ORKID Bundled Intervention
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Renal Recovery
Description: Days after study enrollment before renal recovery, defined as being alive and off dialysis for 14 consecutive days.
Time Frame: Study day 90
Population: Only 1 participant was enrolled in this study, due to the possibility of identification, data will not be presented.
Arm/Group | ORKID Bundled Intervention
Number analyzed (Participants) | 0

5. Secondary Outcome: Proportion of Dialysis Sessions Complicated by Intradialytic Hypotension
Description: Defined as nadir systolic blood pressure < 90 mmHg.
Time Frame: Study day 90
Population: Only 1 participant was enrolled in this study, due to the possibility of identification, data will not be presented.
Arm/Group | ORKID Bundled Intervention
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants Enrolled Per Month
Description: Recruitment rate
Time Frame: Total study duration, anticipated 1 year
Population: Only 1 participant was enrolled in this study, due to the possibility of identification, data will not be presented.
Arm/Group | ORKID Bundled Intervention
Number analyzed (Participants) | 0

7. Secondary Outcome: Ratio of the Number of Participants Who Meet Inclusion Criteria to the Number of Participants Enrolled
Description: Screening-to-recruitment ratio
Time Frame: Total study duration, anticipated 1 year
Population: Only 1 participant was enrolled in this study, due to the possibility of identification, data will not be presented.
Arm/Group | ORKID Bundled Intervention
Number analyzed (Participants) | 0

8. Secondary Outcome: Modified Dialysis Symptom Index Score
Time Frame: Study day 0, 7, 14, 28, and 90
Population: Only 1 participant was enrolled in this study, due to the possibility of identification, data will not be presented.
Arm/Group | ORKID Bundled Intervention
Number analyzed (Participants) | 0

9. Secondary Outcome: Kidney Disease Quality of Life-36 Score
Time Frame: Study day 0, 7, 14, 28, and 90
Population: Only 1 participant was enrolled in this study, due to the possibility of identification, data will not be presented.
Arm/Group | ORKID Bundled Intervention
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 month
Description: Only 1 participant was enrolled in this study, due to the possibility of identification, data will not be presented.
Arm/Group | ORKID Bundled Intervention
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT05158153/Prot_SAP_000.pdf